CLINICAL TRIAL: NCT02837042
Title: Phase II Trial of Pembrolizumab for Advanced Penile Squamous Cell Carcinoma Following Previous Chemotherapy
Brief Title: Trial of Pembrolizumab for Advanced Penile Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lisle Nabell, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F160426013 (UAB 15107)
Record Dates: First submitted 2016-07-01; First posted 2016-07-19 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Penile Squamous Cell Carcinoma
Keywords: penile cancer; Pembrolizumab; penile squamous cell carcinoma; squamous cell cancer
MeSH Terms: conditions — Penile Neoplasms; Neoplasms, Squamous Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab 200 mg (Experimental): Once eligibility is confirmed, the patient will start treatment cycles with Pembrolizumab at 200 mg given intravenously on the first day of each cycle. Each cycle corresponds to a duration of 3 weeks.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously every 3 weeks.
  Other Names: Keytruda

SUMMARY:
Penile squamous cell carcinoma (PSCC) is relatively rare but exhibits higher incidences in less developed countries. PSCC is a highly aggressive malignancy characterized by early spread. Pembrolizumab has recently been FDA-approved for the treatment of melanoma but will serve as the investigational agent for this penile cancer study.

DETAILED DESCRIPTION:
This is a multicenter trial to evaluate Pembrolizumab for patients with advanced penile squamous cell carcinoma following prior chemotherapy. Participating institutions are the University of Alabama at Birmingham (coordinating center), M.D. Anderson Cancer Center, University of Michigan, University of Minnesota, and Emory University. Patients will receive intravenous Pembrolizumab every 3 weeks and undergo a clinical exam. Radiographic scans will be done at baseline and every 9 weeks. Therapy will continue until disease progression or there are intolerable toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced unresectable or metastatic stage 4 (i.e. T4 or N3 or M1) PSCC
2. Radiologic evidence for progressive disease after ≥1 prior chemotherapy regimen
3. Be at least 18 years of age on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
6. Demonstrate adequate organ function with all screening labs being performed within 14 days of treatment initiation.

   * Absolute neutrophil count (ANC) ≥1,500 /microLiters (mcL)
   * Platelets ≥100,000/mcL
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin dependency (within 7 days of assessment)
   * Serum creatinine ≤1.5 X upper limit of normal (ULN); alternately measured or calculated creatinine clearance ≥30 mL/min with creatinine levels >1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl)
   * Serum total bilirubin ≤1.5 X ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels >1.5 ULN
   * Aspartate Transaminase (AST), also known as Serum Glutamic-Oxaloacetic Transaminase (SGOT) and Alanine Aminotransferase (ALT), also known as Serum Glutamic-Pyruvic Transaminase (SGPT) ≤ 2.5 X ULN or ≤ 5 X ULN for subjects with liver metastases
   * Albumin >2.5 mg/dL
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
7. Subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
8. Formalin-fixed paraffin embedded (FFPE) tumor tissue from previous biopsy is requested, but not mandatory.
9. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Hypersensitivity to Pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant expecting to father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-Programmed Cell Death-1 (PD-1), anti-PD-Ligand 1 (L1), or anti-PD-Ligand 2 (L2) agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (HCV) (e.g., HCV RNA [qualitative] is detected).
18. Has known active Tuberculosis infection.
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisle Nabell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Winship Cancer Institute at Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate
Description: The response rate will be evaluated every 3 weeks using the criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in addition to immune related criteria based on patterns of response.
Time Frame: Baseline up to two years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The duration of time from the start of treatment to the first documentation of tumor progression.
Time Frame: Baseline up to two years
Population: Since the trial stopped due to poor accrual, and more censored patients, the 95% CI for median PFS and OS could not be determined. We are reporting median values without CI.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 6
days | 91 [NA to NA] — The study was ended prematurely due to poor accrual and only two patients progressed while the rest were lost to follow up. The statistical analysis will not give a reliable range except median based on two findings

3. Secondary Outcome: Overall Survival
Description: Length of subject survival after starting study treatment
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
Population: Due to poor accrual, low sample size, and higher number of patients censored, the 95% CI for median OS and PFS could not be determined.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 6
days | 307 [NA to NA] — The study was ended prematurely due to poor accrual and only two patients progressed while the rest were lost to follow up. The statistical analysis will not give a reliable range except median based on two findings

4. Secondary Outcome: Number of Patients With Adverse Events
Description: Adverse events reporting will be graded following the National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
Time Frame: Baseline up to two years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants | 4

ADVERSE EVENTS:
Time Frame: From baseline through one year after the end of the study, up to 2 years.
Description: The study was closed prematurely due to poor accrual and substantial loss to follow-up of patients.
Arm/Group | Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=6)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=6)
Fever (Infections and infestations) | 1 (1)
Hyponatremia (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT02837042/Prot_SAP_000.pdf